CLINICAL TRIAL: NCT04770948
Title: A Study Evaluating the Diagnostic Yield and Safety of the 19-GaUge vs 22-Gauge EBUS-TBNA Needle in Subjects With Suspected Sarcoidosis (GUESS)
Brief Title: An RCT of 19G EBUS-TBNA Needle in Suspected Sarcoidosis
Acronym: GUESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: All India Institute of Medical Sciences (Other); Apollo Hospitals Enterprise Limited (Other); Jaipur Golden Hospital, New Delhi (Unknown); Rajiv Gandhi Cancer Institute & Research Center, India (Other); Institute of Pulmonology, Medical Research, and Development, Mumbai (Unknown); All India Institute of Medical Sciences, Bhopal (Other); Asian Institute of Gastroenterology, Hyderabad (Unknown); Yashoda Hospitals, Hyderabad (Unknown); City Clinic and Bhailal Amin General Hospital, Vadodara (Unknown)
Responsible Party: Principal Investigator, Ritesh Agarwal, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SPL822
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 19G (Experimental): 19 gauge EBUS-TBNA needle
  Interventions: Device: 19 gauge needle
- 22G (Active Comparator): 22 gauge EBUS-TBNA needle
  Interventions: Device: 22 gauge needle

INTERVENTIONS:
Device: 19 gauge needle — EBUS-TBNA performed using 19G needle
  Arms: 19G
Device: 22 gauge needle — EBUS-TBNA performed using 22G needle
  Arms: 22G

SUMMARY:
Sarcoidosis is an idiopathic disorder characterized by granulomatous inflammation involving various organ systems. The lung and mediastinal lymph nodes are the most commonly involved structures in sarcoidosis. In the presence of intrathoracic lymph nodes, transbronchial needle aspiration (TBNA) is a useful diagnostic modality, which is now guided using endobronchial ultrasound (EBUS).

We hypothesize that the 19-gauge EBUS-TBNA needle will have a higher yield as compared to the conventional 22-gauge EBUS-TBNA needle in intrathoracic lymphadenopathy due to sarcoidosis. In this study, we plan to evaluate the yield and safety of the 19-gauge needle vs. the conventional 22-gauge EBUS-TBNA needle in patients with sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is an idiopathic disorder characterized by granulomatous inflammation involving various organ systems. The disease is diagnosed based on a suggestive clinicoradiological picture and the presence of non-caseating granulomas in the involved organ, after excluding known causes of granulomatous inflammation. The lung and mediastinal lymph nodes are the most commonly involved structures in sarcoidosis. Various bronchoscopic techniques such as endobronchial biopsy (EBB), transbronchial biopsy (TBLB) and transbronchial needle aspiration (TBNA) are commonly used for acquiring tissue samples.

In the presence of intrathoracic lymph nodes, TBNA is a useful diagnostic modality, especially when combined with endobronchial and transbronchial biopsies. At most centers, TBNA is now guided using endobronchial ultrasound (EBUS). The technique is minimally invasive and also offers the advantage of a selection of the appropriate node for sampling based on the ultrasonographic characteristics. Several studies have demonstrated the superiority of EBUS-TBNA over conventional TBNA (TBNA performed without real-time guidance).

Several technical aspects of EBUS-TBNA have been studied to optimize the yield including the number of aspirations or passes required per lymph node station, needle gauge (21 vs. 22 gauge), suction pressure, the distance travelled by the needle within the lymph node, the number of needle agitations required during a pass, and others.

The novel 19-G Vizishot FLEX EBUS needle (Olympus) is composed of a more flexible material (nitinol) than the 22-G EBUS needle. This allows it to have a larger inner diameter with the same outer diameter as a 22-G EBUS needle. Recent studies have shown that the 19-G needle is safe and has a comparable yield to smaller bore needles. In case of suspected lymphadenopathy due to malignant disorders, aspiration using smaller gauge needles may yield sufficient material for diagnosis. However, in sarcoidosis, larger nodal tissue obtained with a thicker bore needle, the 19-gauge needle, may potentially increase the identification of granulomas. We hypothesize that the 19-gauge EBUS-TBNA needle will have a higher yield as compared to the conventional 22-gauge EBUS-TBNA needle in intrathoracic lymphadenopathy due to sarcoidosis. In this study, we plan to evaluate the yield and safety of the 19-gauge needle vs. the conventional 22-gauge EBUS-TBNA needle in patients with sarcoidosis.

ELIGIBILITY:
Inclusion Criteria: All the following

* Age at least 18 years
* Clinicoradiological suspicion of sarcoidosis where EBUS-TBNA is being planned
* Enlarged bilateral hilar and/or mediastinal lymph nodes >10 mm (any axis) on computed tomography of the chest
* Ability to provide informed consent to participate in the study.

Exclusion Criteria: Patients with any of the following will be excluded

* Asymmetric lymph nodes
* Lymph nodes with significant hypodense areas suggestive of necrosis
* Tuberculin skin test >10 mm
* Hypoxemia (SpO2 <92% on FiO2 of 0.3)
* Treatment with systemic glucocorticoids for >2 weeks in the preceding three months
* Diagnosis of sarcoidosis possible with another minimally invasive technique such as skin biopsy or peripheral lymph node biopsy
* Failure to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of EBUS-TBNA samples | 6 months
  Specimen showing epithelioid cell granulomas or collection of epithelioid cells with a giant cell (or asteroid body or Schaumann body).

SECONDARY OUTCOMES:
Adequacy of EBUS-TBNA samples | 7 days
  Specimen shows a preponderance of lymphocytes or is diagnostic
Complication rate | 7 days
  Complication associated with EBUS-TBNA procedure
Cough visual analog scale (VAS) | 1 day
  Operator-rated visual analog scale (VAS) score for the intensity of subject's cough
Operator VAS | 1 day
  VAS score for ease of performance of the needle puncture and aspiration rated by the operator

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided